CLINICAL TRIAL: NCT05993442
Title: Optimising Kangaroo Care to Reduce Neonatal Severe Infection/Sepsis and Resistant Bacterial Colonisation Among High-risk Infants in Neonatal Intensive Care: a Pragmatic, Multicentre, Parallel Cluster Randomised Hybrid Implementation-effectiveness Study.
Brief Title: Optimising Kangaroo Care to Reduce Neonatal Severe Infection/Sepsis and Resistant Bacterial Colonisation Among High-risk Infants in NICU.
Acronym: NeoDeco
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: St George's, University of London (Other); European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other); University of Zurich (Other); Universiteit Antwerpen (Other); Charite University, Berlin, Germany (Other); UMC Utrecht (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NeoDeco
Record Dates: First submitted 2023-06-28; First posted 2023-08-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infection, Bacterial
Keywords: Nosocomial Infection; Prevention; Bacterial; Cluster; Implementation science; Surveillance; Neonatal unit
MeSH Terms: conditions — Bacterial Infections; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimised kangaroo care (Experimental): The sites randomised in this group will adapt the study intervention consisting of:
  Component 1: Skin-to-skin contact for optimised KC, describes the targeted level of early, repeated and sustained skin-to-skin contact (StSC) considered to represent optimised KC in a high-technology neonatal unit environment in which KC is already offered as part of routine care.
  Component 2: Implementation Support aims to engage clinical staff in the neonatal unit who are involved in implementing StSC as part of optimised KC.
  Interventions: Behavioral: Optimised kangaroo care
- Standard of Care (No Intervention): The sites randomised in this group will follow the standard care, including KC and StSC sessions, treatment of severe infections/sepsis and infection prevention and control measures based on current routine local practice. Standard care in all participating NICUs already includes KC but without specific activities to ensure this is implemented according to international best practice recommendations.

INTERVENTIONS:
Behavioral: Optimised kangaroo care — The intervention of optimised KC implementation consists of two components. Component 1 defines the targeted StSC for optimised KC, while component 2 is the implementation support to put in place a tailored implementation strategy.,
  Arms: Optimised kangaroo care

SUMMARY:
NeoDeco is a pragmatic, multicenter, parallel group, cluster randomised hybrid effectiveness-implementation study with baseline assessment, wash-in period and staggered randomisation. All sites will be offered the implementation support for optimised Kangaroo Care (KC) as part of the study; however, intervention sites will be randomised to immediate receipt of implementation support whereas standard care sites will be offered this after the study period.

DETAILED DESCRIPTION:
The NeoDECO trial is a cluster-randomized trial involving up to 24 neonatal units across 5 European countries: Switzerland, Italy, Greece, Spain, and the United Kingdom.

Sites will be grouped into two staggered phases (with at least 10 sites in each). Within each stagger, sites will be randomized to either the intervention arm or the control arm (standard care). Randomisation will occur at the end of the baseline period, which will be identical for all sites. Intervention sites will then undergo a 2-month wash-in phase during which they will receive training and workshops on implementation strategies for optimized Kangaroo Care (KC). Each neonatal unit/site constitutes a cluster, and the intervention is applied at the unit level.

Following the wash-in phase, the intervention period for intervention sites will last 10 months. During this time, optimised KC-defined as early, repeated, and sustained skin-to-skin contact-will be continuously implemented.

All sites, regardless of their allocation (intervention or control arm), will conduct a baseline data collection phase involving clinical surveillance and colonisation assessments. This includes data and sample collection for all consented high-risk babies present in the unit on the day of assessment. Specifically, all sites will collect stool samples weekly during the baseline period and monthly during the wash-in and intervention periods from all high-risk babies present in the unit on the day of the assessment.

Additionally, one representative site per country from the intervention arm will be selected for further in-depth engagement and data collection by the implementation team. This will gather additional information on intervention fidelity and implementation strategies, including acceptability, appropriateness, feasibility, and sustainability.

At the end of the intervention period, all control sites will be supported and trained to implement the optimised KC using the selected implementation strategies.

ELIGIBILITY:
In NeoDeco there are no participant inclusion or exclusion criteria because this is a cluster randomised trial, so the intervention will be applied to all babies admitted to the neonatal intensive care unit as a cluster.

However, the neonatal intensive care units will have to meet the following criteria to be involved in the study:

Inclusion Criteria:

* European NICUs that provide routine care of extremely premature infants (< 28 weeks' gestational age).
* Minimum number of 12 beds offering highest level of neonatal intensive care.
* Availability of or access to -70 to -80°C freezer for storage of research samples.
* Willing to implement optimised KC if allocated to the intervention group.
* Willing to commit to offering the minimum expected target duration or an increase of 50% if NICU is already offering the minimum expected target duration, if allocated to the intervention arm.
* Prepared to implement NeoIPC surveillance
* Adequate resources and expertise and approvals from relevant Research Ethics Committees, as appropriate.

Exclusion Criteria:

* NICU already practices 'long-term' StSC of > 18 hours. Major expected changes in resistant bacterial colonisation pressure during the study period, for example due to planned move to a new ward.
* Participation in other interventional IPC research projects which might directly influence the study intervention or outcome.

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3080 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Neonatal severe infection/sepsis | 12 months
  The cumulative incidence of neonatal severe infection/sepsis in high-risk infants during their NICU stay will be analysed using mixed-effects logistic regression analysis with a random intercept for hospital. The determinant of interest will be the randomly allocated intervention. Co-variates in the analysis include the variables used for restricted randomisation and important individual-level infant characteristics present at admission: birth weight group, gestational age group and mode of delivery (vaginal birth or Caesarean section).
Resistant bacterial colonisation over time | 12 months
  The prevalence of resistant bacterial colonisation over time in high-risk infants admitted to the NICU will be analysed using mixed effects time-series analysis with a random intercept and random time-slope at the hospital level. Individual data will be analysed with a binary outcome (detection or no detection). Data of the pre-trial and full trial period will be visualised, but only PPS collected after the wash-in period (or after the same period in control hospitals) will be analysed in the primary analysis. The two determinants of interest are (1) allocated intervention group and (2) time in months since end of the wash-in period (being zero for control hospitals), including the same co-variates as for neonatal severe infection/sepsis.

SECONDARY OUTCOMES:
Incidence of neonatal sever infections | 12 months
  The study will assess the effect of the intervention among all infants on the cumulative incidence of neonatal severe infection/sepsis, laboratory-confirmed bloodstream infections, clinical sepsis and necrotising enterocolitis (NEC)
Incidence of neonatal morbidity | 12 months
  The study will evaluate the composite outcome of major neonatal morbidity, defined as laboratory-confirmed sepsis, NEC, high-grade ROP, high-grade IVH, BPD or death during NICU stay, and the effect of the intervention in high-risk infants using a negative binomial model, adjusted for the cumulative incidence of the same endpoints in the year before start of the trial.

OTHER OUTCOMES:
Incidence of SSIs | 12 months
  The study will explore the effect of the intervention among high-risk infants and all infants on cumulative incidences of SSIs, including superficial, deep or organ-space SSI, pneumonia (including VAP) and DAIs.
Prevalence of breastfeeding | 12 months
  The study will compare prevalence of breastfeeding and mother's milk intake over time as well as human milk intake among high-risk infants and all infants in both groups.
Incremental cost-effectiveness ratio (ICER) | 12 months
  The incremental cost-effectiveness ratio (ICER) of the intervention compared to the standard care using indicators from the trial outcomes will be calculated to estimate a range of ICERs, including the incremental cost per case of infection averted, cost per life-year gained, and cost per disability-adjusted life-years (DALYs) averted.
Budget impact of the intervention arm | 12 months
  A sensitivity analysis to assess the robustness of cost-effectiveness analyses results to changes in assumptions or inputs will be performed. This may entail testing various scenarios or different assumptions about the costs or benefits of optimised KC. Further, the budget impact of scaling-up the intervention's coverage for the health systems of the countries included in the study will be estimated, if proved effective and cost-effective.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bielicki, PhD, Study Chair — St George's, University of London
Locations (10):
- Greece (5):
  - University General Hospital Attikon, Attiki
  - University Hospital of Heraklion, Heraklion
  - Ioannina University Hospital, Ioannina
  - Hippokration Hospital - Thessaloniki, Thessaloniki
  - Papageorgiou Hospital, Thessaloniki
- Switzerland (5):
  - University of Basel Children's Hospital, Basel
  - Inselspital - University Hospital of Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Children's Hospital of Eastern Switzerland St.Gallen, Sankt Gallen
  - Universitätsspital Zürich - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NeoDeco study is part of the NeoIPC project funded by the European Commission. — https://neoipc.org/